CLINICAL TRIAL: NCT07300774
Title: Transcutaneous Vagus Nerve Stimulation in Premature Ejaculation
Brief Title: Vagus Nerve Stimulation in Premature Ejaculation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Asst. Prof., Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVU00011
Record Dates: First submitted 2025-12-04; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Premature Ejaculation
Keywords: Vagus nerve stimulation; Heart Rate Variability; Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Intervention Model Description: A comparison between transcutaneous auricular vagus nerve stimulation and sham stimulation will be performed.
Who Masked: Outcomes Assessor
Masking Description: In this study, assessor blinding will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation Group (Active Comparator): Transcutaneous auricular vagus nerve stimulation
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Sham Stimulation Group (Placebo Comparator): Sham Stimulation
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Non-invasive electrical stimulation of the vagus nerve via the tragus and conchae

SUMMARY:
Introduction: Premature ejaculation (PE), one of the most common sexual dysfunctions in men, negatively affects sexual function and quality of life. Transcutaneous auricular vagal nerve stimulation (taVNS) provides autonomic regulation non-invasively by balancing the sympathetic and parasympathetic systems.

Objective: To investigate the effectiveness of taVNS on autonomic and sexual function in men with PE and to compare the effectiveness of different taVNS application methods.

Materials and Methods: This prospective, randomized, sham-controlled, single-blind (evaluator) study will be conducted on 102 men with PE. Physical, sociodemographic, and clinical characteristics will be evaluated. Heart rate variability will be assessed using the Polar H7 device, premature ejaculation status using the Premature Ejaculation Assessment Questionnaire, and sexual function using the International Index of Erectile Function. Participants will be randomized into two groups (intra-auricular taVNS and sham-taVNS). taVNS treatment will be administered to each group three days per week, with 20-minute sessions, for 12 weeks. For in-ear taVNS, bilateral ear sets with a 36-square-millimeter surface area will be used to stimulate the tragus and concha will be used to stimulate the tragus and concha for intra-auricular taVNS, while adhesive electrode pads with a similar surface area of 36 square millimeters (3 mm × 12 mm) will be used for retroauricular taVNS. The taVNS protocol includes bilateral auricular stimulation for 20 minutes, a stimulation frequency of 25 hertz (Hz), a pulse width of 250 μs, suprathreshold current (0.13-50 mA), and a biphasic mode. Sham groups will also have the same specially designed electrodes placed inside the ear. The device will be turned on but set to 0 mA amplitude, so no electrical stimulation will be delivered.

DETAILED DESCRIPTION:
Premature ejaculation (PE) is one of the most common sexual dysfunctions in men, profoundly affecting the quality of life of both the patient and their partner. Many of the proposed definitions for PE are not based on scientific data and lack diagnostic criteria. The International Society for Sexual Medicine (ISSM) defines PE (lifelong and acquired) as characterized by the following criteria: Ejaculation that occurs almost always or always before or within 1 minute of vaginal penetration (lifelong PE) or a clinically significant decrease in ejaculation latency time, typically to 3 minutes or less (acquired PE); Inability to delay ejaculation in almost all or all vaginal penetrations (lifelong and acquired PE); Negative personal consequences such as distress, anxiety, disappointment, and/or avoidance of sexual intimacy (lifelong and acquired PE). Epidemiological studies based on patient-reported outcome measures have found the prevalence of PE complaints in the male population to be as high as 20-30%. A review of the literature reveals that approaches such as behavioral therapy, exercise programs, neuromuscular electrical stimulation, and yoga are used in the treatment of premature ejaculation, in addition to pharmacological treatment. However, no study has been found that examines the effectiveness of transcutaneous auricular vagal nerve stimulation on autonomic function and PE in men with PE. Therefore, this study was designed to examine the effects of taVNS on autonomic function and PE in men with PE. Participants will be randomly assigned to four groups (intra-auricular taVNS, retro-auricular taVNS, intra-auricular sham-taVNS, and retro-auricular sham-taVNS). The taVNS will be administered to each group three days per week, with 20-minute session durations, for 12 weeks. The taVNS protocol includes bilateral auricular stimulation for 20 minutes, a stimulation frequency of 25 hertz (Hz), a pulse width of 250 μs, suprathreshold current (0.13-50 mA), and a biphasic mode. For intra-auricular taVNS, bilateral ear sets with a 36-square-millimeter surface area to stimulate the tragus and concha will be used for intra-auricular taVNS, and adhesive electrode pads with a similar surface area of 36 square millimeters (3 mm × 12 mm) will be used for retroauricular taVNS. Sham groups will also have the same specially designed electrodes placed intra-auricularly and retroauricularly. The device will be turned on but set to 0 mA amplitude, so no electrical stimulation will occur. Heart rate variability, Premature Ejaculation Assessment Questionnaire, International Index of Erectile Function will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of premature ejaculation according to the International Society for Sexual Medicine (ISSM),
* Having the same, non-pregnant, sexually active partner for at least 6 months,
* Being in a stable, heterosexual relationship,
* Suffering from PE and seeking medical treatment.

Exclusion Criteria:

* Having acquired PE,
* History of vagotomy,
* Having diabetes, hypertension, cardiovascular disease,
* Abnormal neurological examination findings,
* Use of drugs that impair heart rate variability (agents, a-receptor agonists or antagonists, tricyclic or serotonergic antidepressants, antihypertensive drugs)
* History of pelvic surgery,
* Tobacco or alcohol use,
* Any organic cause of PE (as assessed by prostatic secretion analysis, thyroid-stimulating hormone);
* Having a psychiatric disorder,
* Having skin irritation/lesion at the application site,
* International Index of Erectile Function score below 26

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men who experience premature ejaculation will be included in the study.
Enrollment: 102 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | Baseline and at the end of the 12th week
  Heart rate variability will be measured for 5 minutes over the chest using the Polar H7 device.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Cihad Yılmaz, Ph.D., Study Director — Igdir University
Locations (1):
- Bahcesehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A decision on this matter will be made later.

REFERENCES:
- [Background] Ventus D, Jern P. Lifestyle Factors and Premature Ejaculation: Are Physical Exercise, Alcohol Consumption, and Body Mass Index Associated With Premature Ejaculation and Comorbid Erectile Problems? J Sex Med. 2016 Oct;13(10):1482-7. doi: 10.1016/j.jsxm.2016.08.007. Epub 2016 Aug 31. PMID 27590186
- [Background] Jiang M, Yan G, Deng H, Liang H, Lin Y, Zhang X. The efficacy of regular penis-root masturbation, versus Kegel exercise in the treatment of primary premature ejaculation: A quasi-randomised controlled trial. Andrologia. 2020 Feb;52(1):e13473. doi: 10.1111/and.13473. Epub 2019 Nov 20. PMID 31746051
- [Background] La Pera G. Awareness and timing of pelvic floor muscle contraction, pelvic exercises and rehabilitation of pelvic floor in lifelong premature ejaculation: 5 years experience. Arch Ital Urol Androl. 2014 Jun 30;86(2):123-5. doi: 10.4081/aiua.2014.2.123. PMID 25017593